CLINICAL TRIAL: NCT03224117
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Dose Finding Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of DWJ211 in Patient With Moderate or Severe Submental Fat
Brief Title: Clinicial Trial to Evaluate the Efficacy and Safety of DWJ211 in Patient With Moderate or Severe Submental Fat
Acronym: SMF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWJ211001
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Treatment for Submental Fat
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): SQ injection
  Interventions: Drug: Normal saline
- DWJ211_0.5% (Experimental): SQ injection with DWJ211 0.5%
  Interventions: Drug: DWJ211
- DWJ211_1% (Experimental): SQ injection with DWJ211 1.0%
  Interventions: Drug: DWJ211
- DWJ211_2% (Experimental): SQ injection with DWJ211 2.0%
  Interventions: Drug: DWJ211

INTERVENTIONS:
Drug: DWJ211 — inject the Drug into submental fat via subcutaneous
  Arms: DWJ211_0.5%; DWJ211_1%; DWJ211_2%
Drug: Normal saline — inject the Drug into submental fat via subcutaneous
  Arms: Placebo

SUMMARY:
evaluate the efficacy and safety of DWJ211 in patient with moderate or severe submental fat

DETAILED DESCRIPTION:
DWJ211

_ reduction of moderate or severe submental fat

ELIGIBILITY:
Inclusion Criteria:

1. submental fat grade by the investigator as 2 or 3 using the PA-SMFRS and graded by the subject as 2 or 3 using the SA-SMFRS as determined on Visit 1.
2. Dissatisfaction with the submental area expressed by the subject as a rating of 1~3 using the SSS as determinded on Visit 1.
3. less than 35kg/m2 in body mass index on Visit1.
4. subject who will agree with the no treatment for the procedure that may affect to reduction or the submental fat.
5. subject who will agree with maintaining their body weight.

Exclusion Criteria:

1. History of any intervention to treat SMF
2. History of trauma associated with the chin or neck areas that in the judgement of the investigator may affect evaluation of safety or efficacy of treatment.
3. Evidence of any cause of enlargement in the submental area.
4. history or current symptoms of dysphagia.
5. a result on coagulation tests that indicates the presence of any clinically significant bleeding disorder.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
2-grade response : PA-SMFRS | 4 week after last treatment
  proportion of subject who simultaneously have at least a 2 grade improvement from baseline on the PA-SMFRS at 4weeks after the last treatment
2-grade response : SA-SMFRS | 4 week after last treatment
  proportion of subject who simultaneously have at least a 2-grade improvement from baseline on the SA-SMFRS at 4weeks after the last treatment
1-grade response : PA-SMFRS | 4 week after last treatment
  proportion of subject who simultaneously have at least a 1-grade improvement from baseline on the PA-SMFRS at 4weeks after the last treatment
1-grade response : SA-SMFRS | 4 week after last treatment
  proportion of subject who simultaneously have at least a 1-grade improvement from baseline on the SA-SMFRS at 4weeks after the last treatment

SECONDARY OUTCOMES:
MRI volume response rate | 4 week after last treatment
  change rate of reduction in SMF volume
improvement: SA-SMFIS | 4 week after last treatment
  improvement in the Subject reported submental fat impact scale overall score
obtained 5 score : SSS | 4 week after last treatment
  proportion of subjects who have more than 5 score on the SSS(somewhat satisfied)
thickness response rate : caliper | 4 week after last treatment
  change rate of reduction in SMF volume

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, MD, PhD, Study Chair — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Yang-won Lee, MD, PhD, Principal Investigator — Konkuk University Medical Center; Chong-hyun Won, MD, PhD, Principal Investigator — Seoul Asan medical center
Locations (3):
- South Korea (3):
  - Chung-ang university hospital, Seoul
  - Konkuk university medical center, Seoul
  - Seoul Asan medical center, Seoul

IPD SHARING:
Plan to Share IPD: No